CLINICAL TRIAL: NCT00857688
Title: Randomized Clinical Study to Evaluate the Effectiveness and Safety of the Drug Topic Bismu-Jet ® (Bismuth Tartrate, Neomycin Sulphate and Procaine Hydrochloride) Compared to Placebo in Improvement of Signs and Symptoms of Ulcerations Caused Disease.
Brief Title: Efficacy of the Combination Bismuth + Neomycin + Procaine in the Treatment of Recurrent Aphthous Ulceration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre FRederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BNPEMS0209
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Aphtous Ulcers
Keywords: aphtous; bismuth; procain; neomycin; Efficacy of the Association in Treatment of Aphtous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Test (Experimental): Patients will recieve the association.
  Interventions: Drug: Bismu-Jet
- 2 (Placebo Comparator): Placebo: Menthol, saccharin sodium, propylene glycol, sodium hydroxide, glycerol, ethyl alcohol, water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bismu-Jet — Bismuth sodium tartrate, neomycin sulfate, procain hydrocloride
  Arms: 1 - Test
Other: Placebo — Placebo: Menthol, saccharin sodium, propylene glycol, sodium hydroxide, glycerol, ethyl alcohol, water
  Arms: 2

SUMMARY:
To evaluate the efficacy of the product Bismu-Jet ® (bismuth tartrate and sodium, neomycin sulfate and procaine hydrochloride) produced by EMS S / A compared to placebo in reducing the signs and symptoms resulting from UAR in patients of both sexes, with age over 12 years.

DETAILED DESCRIPTION:
The period of practical study will be conducted at the Center for Orofacial Rehabilitation Aesthetics, located in Campinas-SP, where there are several beds and a large number of people served by dentists attending post-graduate, under the supervision of Dr. Claudio Azenha. Thus, patients are instructed to find the center if they experience the first signs of UARs.

Will be included only where the top of the table has not extrapolated 48 hours. These patients will be referred to the visit of screening and early treatment (day 0 - Visit 01). At a screening visit will be informed all the relevant aspects of research, enabling the patient judge the feasibility of their participation in the study. After signing the Informed Consent, patients will be randomized and will receive one of the treatments. This consultation will be a clinical examination where the examiner will tell the lesions and measure the size of each. Besides the clinical examination there is a subjective test, in which the patient must consider the intensity of pain you're feeling at that moment, using the visual analogue scale (VAS). The drug will be administered by the investigator, the patient showing the correct way of administration. After 15 minutes, the pain will be measured again, using the VAS.

After three days, patients should return for the 02 tour, which will be clinically evaluated and will be assessed for intensity of pain, in addition to the reporting of adverse events. The same procedures will be repeated in the return of seven days (Visit 03). This visit some patients may receive high clinic.

The study will be finalized after 14 days of treatment (Visit 04), when patients must return to the office to the final evaluations, as will high or be exempted from the clinical study.

Patients who do not have improvement in time, receive replacement therapy funded by the sponsor and provided by waxen, according to the needs of each individual case, judged by expert researchers.

ELIGIBILITY:
Inclusion Criteria:

* Consistency with the purposes of the study and all topics of FICT;
* Age above 12 years;
* Both sexes;
* Diagnosis of type UAR minor

Exclusion Criteria:

* Use of nutritional supplements such as iron, folic acid and vitamins of the B complex;
* immunocompromised;
* systemic diseases (endocrine-metabolic);
* rheumatic diseases;
* Pregnancy and lactation;
* Use of topical or systemic corticosteroids;
* UAR type major;
* UAR type Herpetiformis;
* UAR over 48 hours of development;
* Background allergic to any components of the formula.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The pain will be assessed by visual analogue scale. Will evaluate the size of the lesion using a ruler created specifically for this study The number of lesions will be evaluated by counting. | V0 - 1st day, V1 - 3st day, V2 - 7th day, V3 - 14th day

SECONDARY OUTCOMES:
safety will be assessed by the incidence of adverse reactions | V0 - 1st day, V1 - 3st day, V2 - 7th day, V3 - 14th day

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil